CLINICAL TRIAL: NCT06970782
Title: A Randomized, Controlled, Open Label, Multicenter Phase III Study to Evaluate the Efficacy and Safety of Vebreltinib in Combination With PLB1004 Versus Platinum-based Doublet Chemotherapy in Patients With EGFR Mutations, MET Amplification and/or Overexpression, Locally Advanced or Metastatic Non-Small Cell Lung Cancer Following EGFR-TKI Treatment Failure
Brief Title: Vebreltinib Plus PLB1004 Versus Platinum-based Doublet Chemotherapy in Patients With EGFRm, MET+, Locally Advanced or Metastatic NSCLC Following EGFR-TKI Failure
Acronym: KYLIN-3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLB1001/PLB1004-NSCLC-III-01
Record Dates: First submitted 2025-04-25; First posted 2025-05-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: NSCLC; Lung Cancer; MET Amplification; EGFR L858R; EGFR Exon 19 Deletion; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vebreltinib 150mg BID plus PLB1004 80mg QD (Experimental): Subjects will receive Vebreltinib 150mg orally twice per day (BID) plus PLB1004 80mg orally once per day (QD),21day cycles until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
  Interventions: Drug: Vebreltinib; Drug: PLB1004
- Pemetrexed plus cisplatin/carboplatin (Active Comparator): Subjects randomized to the control group will receive pemetrexed 500 mg/m² + platinum-based chemotherapy (carboplatin AUC 5 or cisplatin 75 mg/m²) via intravenous infusion for 4-6 cycles (determined by the investigator) as initial therapy, followed by pemetrexed maintenance therapy (500 mg/m²) until disease progression, intolerable toxicity, initiation of new antitumor therapy, death, loss to follow-up, or other treatment-terminating conditions (whichever occurred first)
  Interventions: Drug: Pemetrexed plus Carboplatin or Cisplatin

INTERVENTIONS:
Drug: Vebreltinib — Subjects will receive Vebreltinib Enteric-coated Capsule orally twice per day (BID).
  Other Names: Bozitinib; PLB1001
  Arms: Vebreltinib 150mg BID plus PLB1004 80mg QD
Drug: PLB1004 — Subjects will receive PLB1004 80mg orally once per day (QD).
  Other Names: Andamertinib
  Arms: Vebreltinib 150mg BID plus PLB1004 80mg QD
Drug: Pemetrexed plus Carboplatin or Cisplatin — Subjects randomized to the control group received pemetrexed 500 mg/m² + platinum-based chemotherapy (carboplatin AUC 5 or cisplatin 75 mg/m²) via intravenous infusion for 4-6 cycles (determined by the investigator) as initial therapy, followed by pemetrexed maintenance therapy (500 mg/m²) until disease progression, intolerable toxicity, initiation of new antitumor therapy, death, loss to follow-up, or other treatment-terminating conditions (whichever occurred first).
  Arms: Pemetrexed plus cisplatin/carboplatin

SUMMARY:
Efficacy and Safety of Vebreltinib in Combination With PLB1004 Versus Platinum-based Doublet Chemotherapy in Patients With EGFR Mutations, MET Amplification and/or Overexpression, Locally Advanced or Metastatic Non-Small Cell Lung Cancer Following EGFR-TKI Treatment Failure

DETAILED DESCRIPTION:
A Randomized, Controlled, Open Label, Multicenter Phase III Study to Evaluate the Efficacy and Safety of Vebreltinib in Combination With PLB1004 Versus Platinum-based Doublet Chemotherapy in Patients With EGFR Mutations, MET Amplification and/or Overexpression, Locally Advanced or Metastatic Non-Small Cell Lung Cancer Following EGFR-TKI Treatment Failure

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Aged at least 18 years old.
3. Histologically or cytologically confirmed locally advanced or metastatic NSCLC (stage IIIB~IV).
4. At least one measurable lesion as defined by RECIST V1.1.
5. ECOG performance status 0 to 1.

Exclusion Criteria:

1. There are mutations of ALK or ROS1.
2. Have symptomatic and neurologically unstable central nervous system (CNS) metastases or CNS disease that requires increased steroid doses for control.
3. Before randomization, patients did not recover from any toxicity and/ or complications of previous chemotherapy, surgery, radiotherapy and other anti-cancer treatments, that is, did not fall to grade 1 or lower (National Cancer Research Common Toxicity Criteria for Adverse Events [NCI-CTCAE] v5.0), except for hair loss and irrecoverable permanent radiation damage.
4. Major surgery or had significant traumatic injury within 4 weeks prior to the first dose of the investigational product.
5. Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) by BICR | 2 years
  Progression-free survival (PFS) as assessed by a Blind Independent Center Review Committee (BICR) with reference to RECIST v1.1 for Solid tumors.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) by the investigator | 2 years
  Refer to RECIST v1.1, PFS assessed by the investigator.
The objective response rate of the tumor (ORR) | 2 years
  Refer to RECIST v1.1, ORR assessed by the investigator and BICR.
Duration of Response (DoR) | 2 years
  Refer to RECIST v1.1, DoR assessed by the investigator and BICR.
The disease control rate (DCR) | 2 years
  Refer to RECIST v1.1, DCR assessed by the investigator and BICR.
Overall Survival (OS) | 3 years
  OS is defined as the time from the date of the first dose until the date of death due to any cause.
Objective Response Rate (ORR) in subjects with baseline intracranial metastases | 2 years
  Refer to RECIST v1.1，ORR assessed by the investigator and BICR.
The Disease Control Rate (DCR) in subjects with baseline intracranial metastases | 2 years
  Refer to RECIST v1.1, DCR assessed by the investigator and BICR.
Duration of Response (DoR) in subjects with baseline intracranial metastases | 2 years
  Refer to RECIST v1.1, DoR assessed by the investigator and BICR.
Progression-Free Survival (PFS) in subjects with baseline intracranial metastases | 2 years
  Refer to RECIST v1.1, PFS assessed by the investigator and BICR.
Incidence of Treatment-Emergent Adverse Events | 2 years
  Incidence of Treatment-Emergent Adverse Events (TEAEs),A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Plasma concentrations of Vebreltinib and PLB1004 | 2 years
  Plasma concentrations of Vebreltinib and PLB1004.
Second progression-free survival (PFS2) | 2 years
  Investigator-assessed second progression-free survival (PFS2).
Assess the Quality of Healthy Living About Patients（EQ-5D-5L） | 2 years
  Use the EQ-5D-5L scale to measure patients' quality of healthy living. It has 5 items (Mobility, Self-care, Usual activities, Pain/discomfort, Depression/anxiety). Each item contains 5 levels: 1= no difficulty, 2= slight difficulty, 3= moderate difficulty, 4= serious difficulty, 5= extremely serious difficulty. The higher the score has the worse the health.
  Then, the score calculation of the European Five-Dimensional Health Scale is based on the calculation formula published by the EuroQol Group. Based on 5 combinations of different severity levels, a score of 0 to 1 is obtained. 0 is the least healthy and 1 is the most healthy.

IPD SHARING:
Plan to Share IPD: No